CLINICAL TRIAL: NCT05478499
Title: A Phase 3B/4, Multicenter, Randomized, Double-blind Placebo-controlled Study to Evaluate the Efficacy and Safety of Deucravacitinib in Participants With Moderate-to-severe Scalp Psoriasis (PSORIATYK SCALP)
Brief Title: Efficacy and Safety of Deucravacitinib Versus Placebo in Participants With Moderate-to-severe Scalp Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM011-220; 2022-000797-26 (EudraCT Number); U1111-1274-7417 (Registry Identifier: WHO)
Record Dates: First submitted 2022-07-27; First posted 2022-07-28 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis
Keywords: Scalp Psoriasis; BMS-986165; Deucravacitinib; Psoriasis; Psoriasis Special Sites
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Deucravacitinib (Experimental)
  Interventions: Drug: Deucravacitinib
- Placebo then Deucravacitinib (Placebo Comparator)
  Interventions: Drug: Deucravacitinib; Other: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Other Names: BMS-986165
Other: Placebo — Specified dose on specified days
  Arms: Placebo then Deucravacitinib

SUMMARY:
The purpose of this study is to compare the efficacy and safety of deucravacitinib to placebo in participants with moderate-to-severe scalp psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women diagnosed with stable plaque psoriasis with scalp involvement for 6 months or more. Stable psoriasis is defined as no morphology changes or significant flares of disease activity in the opinion of the Investigator
2. Deemed by the Investigator to be a candidate for phototherapy or systemic therapy
3. Moderate-to-severe scalp psoriasis as defined by scalp-specific Physician's Global Assessment (ss-PGA) ≥ 3; ≥ 20% scalp surface area (SSA); Psoriasis Scalp Severity Index (PSSI) ≥ 12 at the Screening visit and Day 1
4. ≥ 3% of Body Surface Area (BSA) involvement at the Screening visit and Day 1
5. Evidence of plaque psoriasis in a non-scalp area
6. Failed to respond to, or intolerant of ≥ 1 topical therapy for scalp psoriasis

Exclusion Criteria:

* Target Disease Exceptions:

  1. Has nonplaque psoriasis (ie, guttate, inverse, pustular, erythrodermic or drug-induced psoriasis) at Screening or Day 1 Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Chair — Bristol-Myers Squibb
Locations (29):
- United States (14):
  - Local Institution - 0001, Hot Springs, Arkansas
  - Local Institution - 0007, Indianapolis, Indiana
  - Local Institution - 0041, Louisville, Kentucky
  - Local Institution - 0022, Rockville, Maryland
  - Local Institution - 0008, Beverly, Massachusetts
  - Local Institution - 0047, Bloomfield Hills, Michigan
  - Local Institution - 0002, New Brighton, Minnesota
  - Local Institution - 0049, East Windsor, New Jersey
  - Local Institution - 0051, Kew Gardens, New York
  - Local Institution - 0003, Portland, Oregon
  - Local Institution - 0005, Pittsburgh, Pennsylvania
  - Local Institution - 0033, Houston, Texas
  - Local Institution - 0004, San Antonio, Texas
  - Local Institution - 0006, Norfolk, Virginia
- France (3):
  - Local Institution - 0019, Paris
  - Local Institution - 0040, Romans-sur-Isère
  - Local Institution - 0044, Rouen
- Germany (5):
  - Local Institution - 0038, Witten, Deutschland
  - Local Institution - 0013, Frankfurt am Main, Hesse
  - Local Institution - 0048, Hamburg
  - Local Institution - 0012, Lübeck
  - Local Institution - 0011, Mahlow
- Poland (4):
  - Local Institution - 0026, Krakow
  - Local Institution - 0017, Lodz
  - Local Institution - 0014, Rzeszów
  - Local Institution - 0015, Wroclaw
- United Kingdom (3):
  - Local Institution - 0031, London, Greater London
  - Local Institution - 0045, Salford, Greater Manchester
  - Local Institution - 0039, Southampton, HAMPSHIRE

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 154 randomized and treated
Groups:
- Deucravacitinib: Deucravacitinib 6 mg daily (QD)
- Placebo: Placebo matching Deucravacitinib daily (QD)
Period: Placebo Controlled: Week 0 - 16
Arm/Group | Deucravacitinib | Placebo
Started (Randomized and treated) | 103 | 51
Completed | 94 | 45
Not Completed | 9 | 6
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other reasons | 0 | 2
Period: Active Treatment: Week 16 - Week 52
Arm/Group | Deucravacitinib | Placebo
Started (All participants switched to open-label Deucravacitinib 6 mg QD through Week 52) | 94 | 45
Completed | 80 | 39
Not Completed | 14 | 6
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lack of Efficacy | 4 | 1
Not completed — Adverse Event | 4 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 1 | 0
Not completed — Non-compliance with protocol | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deucravacitinib | Placebo | Total
Number analyzed (Participants) | 103 | 51 | 154
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.8 (15.70) | 43.2 (13.08) | 42.9 (14.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 20 | 65
  Male | 58 | 31 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 95 | 43 | 138
  Unknown or Not Reported | 2 | 0 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Black or African American | 5 | 2 | 7
  Native Hawaiian or other pacific islander | 0 | 0 | 0
  White | 93 | 47 | 140
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Scalp-specific Physician Global Assessment Score of 0 or 1 (Ss-PGA 0/1) at Week 16
Description: ss-PGA 0/1 response as a percentage of participants with an ss-PGA score of 0 (clear) or 1 (almost clear) with at least a 2-point reduction from baseline at Week 16. Scalp lesions are evaluated in terms of clinical signs of redness, thickness, and scaliness and scored on the following 5-point ss-PGA scale: 0 = absence of disease, 1 = very mild disease, 2 = mild disease, 3 = moderate disease, 4 = severe disease.
Time Frame: Baseline and Week 16
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 103 | 51
Percentage of responders
  Full Analysis Set | 48.5 [38.6 to 58.6] | 13.7 [5.7 to 26.3]
  Patient sub-population (s-PGA ≥ 3): number analyzed (Participants) | 96 | 47
  Patient sub-population (s-PGA ≥ 3) | 50.0 [39.6 to 60.4] | 12.8 [4.8 to 25.7]
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Full Analysis Set; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 6.2, 95% CI 2-sided [2.5 to 15.3] — Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Patient sub-population (s-PGA ≥ 3); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 7.0, 95% CI 2-sided [2.7 to 18.4] — Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Participants With a Psoriasis Scalp Severity Index 90 (PSSI 90) at Week 16
Description: PSSI 90 response as a percentage of participants who achieve at least 90% improvement from baseline in the PSSI score at Week 16. PSSI assesses severity of scalp disease in participants with scalp involvement with a 5-point Likert-type scale on the clinical parameters of erythema, induration, and desquamation. The scores are summed and multiplied by an integer (0 to 6) that represents the area of affected scalp. The PSSI score ranges from 0 to 72 with higher scores indicating more severe symptoms.
Time Frame: Baseline and Week 16
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 103 | 51
Percentage of responders
  Full Analysis Set | 38.8 [29.4 to 48.9] | 2.0 [NA to 10.4] — Insufficient number of participants with events. Lower limit value is "< 0.1"
  Patient sub-population (s-PGA ≥ 3): number analyzed (Participants) | 96 | 47
  Patient sub-population (s-PGA ≥ 3) | 40.6 [30.7 to 51.1] | 2.1 [NA to 11.3] — Insufficient number of participants with events. Lower limit value is "< 0.1"
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Full Analysis Set; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 40.2, 95% CI [4.6 to 352.0] — Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Patient sub-population (s-PGA ≥ 3); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 37.3, 95% CI 2-sided [4.4 to 317.6] — Cochran-Mantel-Haenszel

3. Secondary Outcome: Change From Baseline in Scalp-specific Itch Numerical Rating Scale (NRS) Score at Week 16
Description: Change from baseline in scalp-specific itch numerical rating scale (NRS) score at week 16. The scalp-specific itch NRS is an 11-point horizontal scale anchored at 0 and 10 with 0 representing "no scalp itch" and 10 representing "worst scalp itch imaginable.". Overall severity of a participant's itching from scalp psoriasis is indicated by selecting the number that best describes the worst level of scalp itching within the past 24 hours.
Time Frame: Baseline and Week 16
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 103 | 51
Score on a scale
  Full Analysis Set | -3.2 (2.95) | -0.7 (2.27)
  Patient sub-population (s-PGA ≥ 3): number analyzed (Participants) | 96 | 47
  Patient sub-population (s-PGA ≥ 3) | -3.3 (2.87) | -0.9 (2.29)
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Full Analysis Set; Test type: Superiority; p < 0.0001, analysis of covariance model; Adjusted mean difference = -2.5, 95% CI [-3.3 to -1.6], Standard Error of Mean 0.42 — analysis of covariance model
Statistical Analysis 2: Comparison: Deucravacitinib vs Placebo; Patient sub-population (s-PGA ≥ 3); Test type: Superiority; p < 0.0001, analysis of covariance model; Adjusted mean difference = -2.4, 95% CI 2-sided [-3.3 to -1.5], Standard Error of Mean 0.44 — analysis of covariance model

4. Secondary Outcome: Percentage of Participants With a Static Physician Global Assessment Score of 0 or 1 (s-PGA 0/1) at Week 16
Description: s-PGA 0/1 response as a percentage of participants with an s-PGA score of 0 (clear) or 1 (almost clear) with at least a 2-point reduction from baseline at Week 16. The s-PGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration. The s-PGA measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as clear (0), almost clear (1), mild (2), moderate (3), or severe (4).
Time Frame: Baseline and Week 16
Population: All randomized participants with a s-PGA ≥ 3 at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 96 | 47
Percentage of responders | 51.0 [40.6 to 61.4] | 4.3 [0.5 to 14.5]
Statistical Analysis 1: Comparison: Deucravacitinib vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 23.9, 95% CI 2-sided [5.4 to 105.6] — Cochran-Mantel-Haenszel

5. Secondary Outcome: Number of Participants Experiencing Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment that does not necessarily have a causal relation with this treatment.
Time Frame: From week 0 through week 16
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 103 | 51
Participants | 73 | 26

6. Secondary Outcome: Number of Participants Experiencing Serious Treatment Emergent Adverse Events (TEAEs)
Description: A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From week 0 through week 16
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 103 | 51
Participants | 1 | 1

7. Secondary Outcome: Number of Participants Experiencing Laboratory Test Results of Worst Toxicity Grade
Description: Laboratory test results summary of Worst toxicity grade in SI units for hematology and chemistry using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade 1= mild and asymptomatic; Grade 2= moderate requiring minimal, local or noninvasive intervention; Grade 3= severe or medically significant but not immediately life-threatening; Grade 4= events are usually severe enough to require hospitalization.
Time Frame: Week 0 through Week 16
Population: All treated participants with baseline and post-baseline laboratory assessments
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 103 | 51
Participants
  Basophils (10^9/L) Grade 1-4 | 0 | 0
  Eosinophils (10^9/L) Grade 1 | 4 | 2
  Eosinophils (10^9/L) Grade 2-4 | 0 | 0
  Hemoglobin (g/L) Grade 1 | 5 | 4
  Hemoglobin (g/L) Grade 2 | 1 | 0
  Hemoglobin (g/L) Grade 3 | 0 | 0
  Leukocytes (10^9/L) Grade 1 | 8 | 1
  Leukocytes (10^9/L) Grade 2 | 0 | 1
  Leukocytes (10^9/L) Grade 3-4 | 0 | 0
  Lymphocytes Blood Test (10^9/L) Grade 1 | 1 | 1
  Lymphocytes Blood Test (10^9/L) Grade 2 | 1 | 0
  Lymphocytes Blood Test (10^9/L) Grade 3-4 | 0 | 0
  Lymphocytes Plasma Test (10^9/L) Grade 1 | 1 | 1
  Lymphocytes Plasma Test (10^9/L) Grade 2 | 1 | 0
  Lymphocytes Plasma Test (10^9/L) Grade 3-4 | 0 | 0
  Neutrophils (x10^9/L) Grade 1 | 5 | 2
  Neutrophils (x10^9/L) Grade 2-4 | 0 | 0
  Platelets (10^9/L) Grade 1-4 | 0 | 0
  Alanine Aminotransferase (U/L) Grade 1 | 8 | 8
  Alanine Aminotransferase (U/L) Grade 2 | 0 | 1
  Alanine Aminotransferase (U/L) Grade 3-4 | 0 | 0
  Albumin (g/L) Grade 1-4 | 0 | 0
  Alkaline Phosphatase (U/L) Grade 1 | 1 | 2
  Alkaline Phosphatase (U/L) Grade 2-4 | 0 | 0
  Aspartate Aminotransferase (U/L) Grade 1 | 5 | 5
  Aspartate Aminotransferase (U/L) Grade 2-4 | 0 | 0
  Bilirubin (umol/L) Grade 1: number analyzed (Participants) | 102 | 51
  Bilirubin (umol/L) Grade 1 | 5 | 3
  Bilirubin (umol/L) Grade 2: number analyzed (Participants) | 102 | 51
  Bilirubin (umol/L) Grade 2 | 1 | 0
  Bilirubin (umol/L) Grade 3-4: number analyzed (Participants) | 102 | 51
  Bilirubin (umol/L) Grade 3-4 | 0 | 0
  Calcium (mmol/L) Grade 1 | 1 | 0
  Calcium (mmol/L) Grade 2-4 | 0 | 0
  Chloride (mmol/L) Grade 1-4 | 0 | 0
  Cholesterol (mmol/L) Grade 1: number analyzed (Participants) | 100 | 48
  Cholesterol (mmol/L) Grade 1 | 5 | 0
  Cholesterol (mmol/L) Grade 2-4: number analyzed (Participants) | 100 | 48
  Cholesterol (mmol/L) Grade 2-4 | 0 | 0
  Creatine Kinase (U/L) Grade 1-4: number analyzed (Participants) | 1 | 0
  Creatine Kinase (U/L) Grade 1-4 | 0 |
  Creatinine (umol/L) Grade 1 | 3 | 0
  Creatinine (umol/L) Grade 2 | 1 | 0
  Creatinine (umol/L) Grade 3-4 | 0 | 0
  Direct Bilirubin (umol/L) Grade 1-4: number analyzed (Participants) | 6 | 4
  Direct Bilirubin (umol/L) Grade 1-4 | 0 | 0
  Glucose (mmol/L) Grade 1 | 2 | 0
  Glucose (mmol/L) Grade 2-4 | 0 | 0
  Lactate Dehydrogenase (U/L) Grade 1-4: number analyzed (Participants) | 1 | 0
  Lactate Dehydrogenase (U/L) Grade 1-4 | 0 |
  Magnesium (mmol/L) Grade 1-4: number analyzed (Participants) | 1 | 0
  Magnesium (mmol/L) Grade 1-4 | 0 |
  Phosphate (mmol/L) Grade 1-4 | 0 | 0
  Potassium (mmol/L) Grade 1 | 6 | 2
  Potassium (mmol/L) Grade 2 | 8 | 1
  Potassium (mmol/L) Grade 3 | 0 | 1
  Potassium (mmol/L) Grade 4 | 0 | 0
  Sodium (mmol/L) Grade 1 | 0 | 2
  Sodium (mmol/L) Grade 2 | 1 | 0
  Sodium (mmol/L) Grade 3-4 | 0 | 0
  Triglycerides (mmol/L) Grade 1: number analyzed (Participants) | 100 | 48
  Triglycerides (mmol/L) Grade 1 | 27 | 7
  Triglycerides (mmol/L) Grade 2: number analyzed (Participants) | 100 | 48
  Triglycerides (mmol/L) Grade 2 | 2 | 3
  Triglycerides (mmol/L) Grade 3: number analyzed (Participants) | 100 | 48
  Triglycerides (mmol/L) Grade 3 | 1 | 0
  Triglycerides (mmol/L) Grade 4: number analyzed (Participants) | 100 | 48
  Triglycerides (mmol/L) Grade 4 | 0 | 1
  Urate (umol/L) Grade 1-4: number analyzed (Participants) | 1 | 0
  Urate (umol/L) Grade 1-4 | 0 |
  Urea Nitrogen (mmol/L) Grade 1-4 | 0 | 0

8. Secondary Outcome: Number of Participants Experiencing Laboratory Abnormalities in Potential Drug-Induced Liver Injury Tests
Description: Number of participants with laboratory abnormalities in potential drug-induced liver injury tests.
  ALT=alanine aminotransferase AST=aspartate aminotransferase ULN=upper limit of normal
Time Frame: Week 0 through Week 16
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 103 | 51
Participants
  ALT or AST > 3 X ULN | 0 | 1
  ALT or AST > 5 X ULN | 0 | 0
  Total Bilirubin > 2 X ULN | 0 | 0
  ALT or AST > 3 X ULN and total bilirubin > 2 X ULN on the same day | 0 | 0

9. Secondary Outcome: Number of Participants With Abnormalities in Vital Signs
Description: Number of participants with abnormalities in vital signs including heart rate, systolic blood pressure, and diastolic blood pressure.
Time Frame: Week 0 through Week 16
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib | Placebo
Number analyzed (Participants) | 103 | 51
Participants
  HEART RATE (BEATS/MIN): VALUE > 100 AND CHANGE FROM BASELINE > 30 | 0 | 0
  HEART RATE (BEATS/MIN): VALUE < 55 AND CHANGE FROM BASELINE < -15 | 1 | 3
  HEART RATE (BEATS/MIN): NOT REPORTED | 0 | 0
  SYSTOLIC BLOOD PRESSURE (MMHG): VALUE > 140 AND CHANGE FROM BASELINE > 20 | 3 | 4
  SYSTOLIC BLOOD PRESSURE (MMHG): VALUE < 90 AND CHANGE FROM BASELINE < -20 | 0 | 0
  SYSTOLIC BLOOD PRESSURE (MMHG): NOT REPORTED | 0 | 0
  DIASTOLIC BLOOD PRESSURE (MMHG): VALUE > 90 AND CHANGE FROM BASELINE > 10 | 8 | 3
  DIASTOLIC BLOOD PRESSURE (MMHG): VALUE < 55 AND CHANGE FROM BASELINE < -10 | 0 | 2
  DIASTOLIC BLOOD PRESSURE (MMHG): NOT REPORTED | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their primary data cut-off (Up to 24 months). SAEs and Other AEs were assessed from first dose up to 30 days post last dose (Up to 13 months).
Groups:
- Placebo Controlled - Deucravacitinib; Active Treatment - Deucravacitinib - Deucravacitinib; Active Treatment - Placebo - Deucravacitinib: Deucravacitinib 6 mg daily (QD)
- Placebo Controlled - Placebo: Placebo matching Deucravacitinib daily (QD)
Arm/Group | Placebo Controlled - Deucravacitinib | Placebo Controlled - Placebo | Active Treatment - Deucravacitinib - Deucravacitinib | Active Treatment - Placebo - Deucravacitinib
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/51 | 1/94 | 0/45
Serious Adverse Events (participants affected / at risk) | 1/103 | 1/51 | 4/94 | 0/45
Other Adverse Events (participants affected / at risk) | 47/103 | 14/51 | 42/94 | 16/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Controlled - Deucravacitinib (N=103) | Placebo Controlled - Placebo (N=51) | Active Treatment - Deucravacitinib - Deucravacitinib (N=94) | Active Treatment - Placebo - Deucravacitinib (N=45)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Controlled - Deucravacitinib (N=103) | Placebo Controlled - Placebo (N=51) | Active Treatment - Deucravacitinib - Deucravacitinib (N=94) | Active Treatment - Placebo - Deucravacitinib (N=45)
Acne pustular (Infections and infestations) | 6 | 0 | 3 | 0
COVID-19 (Infections and infestations) | 6 | 4 | 12 | 4
Nasopharyngitis (Infections and infestations) | 16 | 7 | 22 | 8
Upper respiratory tract infection (Infections and infestations) | 12 | 2 | 11 | 3
Headache (Nervous system disorders) | 8 | 2 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 10 | 0 | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 3 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT05478499/Prot_SAP_000.pdf